CLINICAL TRIAL: NCT01736410
Title: A Phase 2 Study of Trastuzumab in Combination With TS-ONE and Cisplatin in Firstline Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Principal Investigator, Choo Su Pin, Doctor, National Cancer Centre, Singapore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC0906
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: HER 2 Positive Advanced Gastric Cancer
MeSH Terms: interventions — Trastuzumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IHC method (Other)
  Interventions: Drug: Trastuzumab, TS ONE, Cisplatin
- FISH method (Other)
  Interventions: Drug: Trastuzumab, TS ONE, Cisplatin

INTERVENTIONS:
Drug: Trastuzumab, TS ONE, Cisplatin — The initial dose of cisplatin is fixed to be 60 mg/m2 and intravenously administered over 1 hour on day 1 of the cycle. TS-ONE is orally administered consecutive 14-day followed by 7-day rest. The initial standard dose of TS-ONE is determined based on the body surface area tabled below. Trastuzumab is intravenously administered with the loading dose of 8 mg/kg followed by HER2-positive advanced GC 21 years or older No prior regimen HER2 protein HER2/neu detection procedure Tissue from (Gastric) Cancer FISH method IHC method negative positive HER-2 negative HER-2 positive Eligible 0 / 1+ 2+ 3+ HER-2 positive Eligible HER-2 negative iii Protocol S1/CDDP/Her V1.3 dated 21 May 10 maintenance dose of 6mg/kg in day 1 of each cycle. The study treatments are repeated every 3 weeks. Study treatment can continue until PD, but cisplatin can be skipped or discontinued if patients experienced unbearable toxicity which comes from cisplatin.

SUMMARY:
To explore overall response rate of trastuzumab combined with TS-ONE based chemotherapy in first-line HER2-positive advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of the stomach and Gastric-esophageal junction.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as more than or equals to 20 mm with conventional techniques or as more than or equals to 10 mm with spiral CT scan.
3. Patients without prior systemic treatment. Patients who completed postoperative adjuvant chemotherapy (and radiotherapy) more than 180 days before may be enrolled.
4. Age more than or equals to 21 years.
5. Life expectancy of greater than 3 months.
6. ECOG performance status less than or equals to 2 (Karnofsky more than or equals to 60%).
7. Patients must have normal organ and marrow function as defined below:

   * Hemoglobin > 8.0 g/dL
   * Leukocytes > 3,000/mcL
   * Absolute neutrophil count > 1,500/mcL
   * Platelets > 100,000/mcL
   * Total bilirubin less than or equals to 1.5 X ULN
   * AST (SGOT)/ALT (SGPT) less than or equals to 3 x institutional upper limit of normal
   * ALP less than or equals to 3 x upper limit of normal*
   * Creatinine within normal institutional limits OR Creatinine clearance** >60 mL/min for patients with creatinine levels above institutional normal

     * In the presence of liver metastasis, patients with AST, ALT and ALP < or = 5 x the upper limit of normal may be admitted. *In the presence of bone metastasis, patients with AST ,ALT and ALP < or = 10x the upper limit of normal maybe admitted. **: Creatinine clearance can be estimated using Cockcroft-Gault formula man: Ccr (mL/min) = body weight (kg) x (140 - age)/(72 x serum creatinine (mg/dL)), woman: Ccr = male Ccr x 0.85]. The above CrCl Formula is to be applied in all sites.
8. Patients who have HER2-positive cancer confirmed with IHC and/or FISH***.

   *** Immunohistochemistry (IHC) for HER-2 is routine as part of pathological evaluation of gastric hybridisation (FISH) for Her2 copy number is required. A copy number value above 2.2 is taken as positive. The sponsors for the drugs used in our investigator initiated trial (Taiho) have kindly agreed to pay for the HER2 FISH test.
9. Patients able to take orally.
10. Patients with left ventricular ejection fraction of at least 50% on MUGA or 2D-echocardiography done within 28 days before enrollment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
11. The effects of proposed regimen on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because antitumor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
12. Ability to understand and the willingness to sign a written informed consent document.
13. Consent for fresh frozen tissue collection, mandatory for patients with primary in-situ tumors and optional for patients without primary in-situ tumors.

    * Tissue collection only applicable to National Cancer Centre (S) and National University Hospital (S)

Exclusion Criteria:

1. Patients who have had radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to treatment administered more than 4 weeks earlier.
2. Patients receiving any other investigational agents.
3. Patients with known brain metastases.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to TS-ONE, cisplatin and trastuzumab or other agents used in the study.
5. Presence of any contraindications to TS-ONE or cisplatin or trastuzumab.
6. Baseline LVEF (Left Ventricular Ejection Fraction) < 50%.
7. Patients with serious (e.g.inpatient care is needed) complications (e.g. intestinal paralysis, intestinal occlusion, interstitial pneumonia or pulmonary fibrosis, poorly-controlled diabetes, renal failure or hepatic cirrhosis).
8. Patients with massive ascites (moderate or higher, beyond the pelvic cavity and retention on the anterior surface of the liver on CT) or massive pleural effusion retention.
9. Patients with fresh bleeding from the digestive tract which needs repeated blood transfusion.
10. Patients with diarrhea (4 or more times per day or watery diarrhea).
11. Previous malignancy other than gastric cancer diagnosed in the last 5 years except for basal cell carcinoma of skin or preinvasive cancer of cervix.
12. Patients with reproductive potential who refuse to use an adequate means of contraception (including male patients).
13. Significant disease or conditions which, in the investigator's opinion, would exclude patient from the study.
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Pregnant or lactating female.
16. HIV-positive patients.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 24 months

SECONDARY OUTCOMES:
Progression free survival (PFS) | 24 months
Overall survival (OS) | 24 months
Time to Treatment Failure (TTF) | 24 months
  Clinical Benefit Rate (CBR), Duration of Response (DR), Safety

CONTACTS AND LOCATIONS:
Overall Officials: Choo Su Pin, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore, Singapore